CLINICAL TRIAL: NCT07240831
Title: Accuracy of a Cuffless Photoplethysmography (PPG) Chest-Patch Monitor for 24-hour Ambulatory Blood Pressure Monitoring
Brief Title: Accuracy of a Cuffless Photoplethysmography (PPG) Chest-Patch Monitor for 24-hour Ambulatory Blood Pressure Monitoring (ABPM)
Acronym: PPG ABPM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biobeat Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Biobeat_CLP_001
Record Dates: First submitted 2025-09-24; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Blood Pressure; Heart Disease; Hypertension (HTN); Blood Pressure Monitoring
Keywords: BLOOD PRESSURE; BLOOD PRESSURE MONITORING; Hypertension (HTN); CUFFLESS PHOTOPLETHYSMOGRAPHY; PPG; CUFFLESS; vital signs
MeSH Terms: conditions — Heart Diseases; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device: Non-invasive monitoring (Experimental): The study is designed as a prospective, multicenter, single arm, validation study that follows the 2023 European Society of Hypertension (ESH) recommendations for the validation of cuffless blood pressure measuring devices.27 There is no primary hypothesis. The study will validate 24-hours blood pressure monitoring using the investigational FDA-cleared device by comparing the level of agreement with parallel measurements obtained by the gold-standard upper arm. The Awake/Asleep test is the first and primary test recommended for this type of device to assess validity.
  Interventions: Device: Model BB-613WP

INTERVENTIONS:
Device: Model BB-613WP — During the study period, participants will undergo standard ABPM monitoring per clinical indication and wear a PPG-based monitor
  Other Names: Biobeat Chest-Patch, PPg-based monitor

SUMMARY:
This study aims to validate the accuracy and reliability of blood pressure (BP) estimates obtained over 24 hours using a PPG-based chest-patch device compared to the gold standard ambulatory blood pressure monitoring (ABPM) method using an upper arm cuff-based oscillometric BP device, in both hypertensive and normotensive individuals referred by their provider to undergo a 24-hours ABPM for clinical indication. The Awake/Asleep test, which is the primary test recommended for automated wearable cuffless BP devices that are cuff-calibrated (based on the 2023 European Society of Hypertension (ESH) recommendations for the validation of cuffless blood pressure measuring devices), will be conducted in this study. The secondary aim of the study is to assess the feasibility and convenience of the PPG-based device.

DETAILED DESCRIPTION:
This study aims to evaluate the accuracy, validity, and efficacy of the Biobeat PPG-based cuffless chest-worn monitor for continuous and ambulatory blood pressure monitoring compared with a standard cuff-based ambulatory blood pressure monitor (ABPM). The study will follow the 2023 European Society of Hypertension (ESH) protocol for validating cuffless BP devices. The Biobeat device is a single-use, wireless, noninvasive patch applied to the chest that continuously measures blood pressure and other vital signs using photoplethysmography (PPG) technology.

The trial is a prospective, multicenter, single-arm validation study in adults undergoing 24-hour ABPM for any clinical indication. Participants will simultaneously wear both the Biobeat device and a standard ABPM for 24 hours. The Biobeat device will be calibrated with three reference cuff measurements at the start of monitoring. Data from both devices will be compared across awake, asleep, and total 24-hour periods to determine agreement in systolic and diastolic blood pressure.

The primary objective is to demonstrate equivalence between the Biobeat PPG-based system and standard ABPM, with accuracy defined as a mean difference ≤5 mmHg and standard deviation ≤8 mmHg. Secondary endpoints include assessment of device performance across different blood pressure ranges and demographic subgroups, as well as participant comfort and usability. The study represents minimal risk to participants; the only potential adverse effect is mild skin irritation from the adhesive patch.

Successful validation will confirm that the Biobeat cuffless PPG-based device provides accurate, reliable 24-hour blood pressure monitoring comparable to existing ABPM systems, supporting its use as a comfortable, patient-friendly alternative for both clinical and ambulatory settings.

ELIGIBILITY:
Inclusion Criteria

* Females and Males subjects 18 years or older (from all skin tones/colors)
* Scheduled for ABPM for hypertension screening, evaluation, or management
* Subjects capable of using an application temporarily downloaded (for the duration of the study) on a personal smart phone device or on a device provided by the study sponsor
* Subjects with Atrial fibrillation or Atrial flutter are eligible to participate if standard cuff-based ABPM monitor can capture blood pressure at initialization

Exclusion Criteria

* Indication for ABPM is orthostatic hypotension or Postural Orthostatic Tachycardiac Syndrome as indicated on the ABPM referral order
* Any neurological, psychological, or other condition impairing the ability to provide informed consent or participate in the study
* Inability to reliably access the Internet via a smart phone
* Not able to perform standard cuff-based ABPM
* Average absolute difference between the two arms is greater than 15 mmHg for Systolic Blood Pressure (SBP) or greater than 10 mmHg Diastolic Blood Pressure (DBP) during the initialization/calibration phase
* Subjects with known allergy to adhesives or skin patches
* Subjects with solid dark tattoos on the area where the PPG-based device is attached
* Subjects who are unwilling to have their chest hair shaved, if needed, to install the device (the device uses adhesives and needs to be in direct contact with the skin without hair)
* Subjects who are unwilling to comply with the study instructions (avoid vigorous exercise and showering for 24 hours while the device is in place)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 24 hours monitoring
  The accuracy and reliability of the PPG-based chest-patch device will be evaluated by comparing its blood pressure measurements with those obtained through the gold-standard upper arm cuff oscillometric ABPM method. Both systolic and diastolic blood pressure values will be assessed.

SECONDARY OUTCOMES:
Secondary Endpoint | 24 hours
  Comparison of the compliance and completeness of the 2 measurement methods. The investigators will report the percentage of participants with at least 30% missed data (defining non-compliance or incomplete study).
Secondary Endpoint | 24 hours
  Convenience of the device (participants' questionnaire) will be assessed.
  Participants will rate the experience on a scale of 1 to 5, with 5 indicating a higher satisfaction score for the following questions:
  1. Comfort level during placement of the monitor
  2. Comfort level during monitoring
  3. Interference with sleep
  4. Interference with daytime activity (i.e., dressing, ambulating, eating)
  5. General satisfaction with the monitoring
     Additional questions-
  6. Which diagnostic option would you recommend to a friend / family member? Options- Biobeat, cuff, either is fine. Answering "Biobeat" will be considered a positive response.
  7. In the future, if you undergo monitoring with Biobeat- how would you prefer to receive the monitor? Options- Mailed directly home, applied at the clinic. Either response is acceptable

OTHER OUTCOMES:
Other Endpoints (exploratory analyses) | 24 hours
  Subgroup analysis based on sex: Sensitivity analyses will assess the agreement between systolic and diastolic blood pressure readings (in mmHg) obtained from the Biobeat wearable monitor and the ABPM. Agreement will be evaluated using descriptive statistics and visual methods (e.g., Bland-Altman plots). No formal statistical subgroup comparisons will be performed
Other Endpoints (exploratory analyses) | 24 hours
  Subgroup analysis based on skin tone: Sensitivity analyses will assess the agreement between systolic and diastolic blood pressure readings (in mmHg) obtained from the Biobeat wearable monitor and the ABPM. Agreement will be evaluated using descriptive statistics and visual methods (e.g., Bland-Altman plots). No formal statistical subgroup comparisons will be performed
Other Endpoints (exploratory analyses) | 24 hours
  Subgroup analysis based on hypertension diagnosis (positive or negative) diagnosed by standard arm-based oscillometric ABPM: Sensitivity analyses will assess the agreement between systolic and diastolic blood pressure readings (in mmHg) obtained from the Biobeat wearable monitor and the ABPM. Agreement will be evaluated using descriptive statistics and visual methods (e.g., Bland-Altman plots). No formal statistical subgroup comparisons will be performed
Other Endpoints (exploratory analyses) | 24 hours
  Subgroup analysis based on participants with atrial fibrillation/atrial flutter: Sensitivity analyses will assess the agreement between systolic and diastolic blood pressure readings (in mmHg) obtained from the Biobeat wearable monitor and the ABPM. Agreement will be evaluated using descriptive statistics and visual methods (e.g., Bland-Altman plots). No formal statistical subgroup comparisons will be performed
Other Endpoints (exploratory analyses) | 24 hours
  Subgroup analysis based on participants with pacemaker: Sensitivity analyses will assess the agreement between systolic and diastolic blood pressure readings (in mmHg) obtained from the Biobeat wearable monitor and the ABPM. Agreement will be evaluated using descriptive statistics and visual methods (e.g., Bland-Altman plots). No formal statistical subgroup comparisons will be performed
Other Endpoints (exploratory analyses) | 24 hours
  Subgroup analysis based on day vs. night analysis: Sensitivity analyses will assess the agreement between systolic and diastolic blood pressure readings (in mmHg) obtained from the Biobeat wearable monitor and the ABPM. Agreement will be evaluated using descriptive statistics and visual methods (e.g., Bland-Altman plots). No formal statistical subgroup comparisons will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Zoghby, M.D., M.B.A., Principal Investigator — Mayo Clinic College of Medicine
Locations (2):
- United States (2):
  - U Health, Miami, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No
This is proprietary company information.